CLINICAL TRIAL: NCT03597607
Title: Efficacy and Cost-Effectiveness of an Intensive and Abbreviated Individualized Smoking Cessation Support Program Delivered by Pharmacists: A Randomized Controlled Trial
Brief Title: Evaluation of an Intensive Individualized Smoking Cessation Program Delivered by Pharmacists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Terri Genge, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREB 6946
Record Dates: First submitted 2017-11-20; First posted 2018-07-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Smoking Cessation; Smoking, Tobacco; Quality of Life
Keywords: Smoking cessation; pharmacist; self-efficacy
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of three groups: intensive smoking cessation program or an abbreviated smoking cessation program.
Who Masked: Outcomes Assessor
Masking Description: Participants will be informed of their group allocation. Health care providers of the intervention will be aware of which program to deliver, therefore knowing group allocation. The investigator will be aware of group allocation. Outcomes will be assessed by a blind data analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Smoking Cessation Group (Experimental): This group will meet with a clinic pharmacist one on one over a period of about 12 weeks. They will have session ranging from 15 mins to 1 hour. Follow-up sessions will occur during quit week(week 1) and at weeks 2, 3, 4, 6, 8, 10, 12 and at 6 months.
  Interventions: Behavioral: Intensive Smoking Cessation Group
- Abbreviated Smoking Cessation Group (Experimental): This group will meet with a clinic pharmacist one on one over a period of about 12 weeks. They will have brief sessions (15-30 mins) at the end of week 1, week 4, week 12 and at 6 months.
  Interventions: Behavioral: Abbreviated Smoking Cessation Group

INTERVENTIONS:
Behavioral: Intensive Smoking Cessation Group — This group will meet with the pharmacist more frequently and for longer periods than other groups.
  Other Names: Intensive group
  Arms: Intensive Smoking Cessation Group
Behavioral: Abbreviated Smoking Cessation Group — This group will meet with the pharmacist less frequently and for shorter periods in comparison to the intensive group.
  Other Names: Abbreviated Group
  Arms: Abbreviated Smoking Cessation Group

SUMMARY:
This study aims to look at the efficacy and impact of a pharmacist-led smoking cessation program. It will assess an intensive program and an abbreviated program, with the latter being evaluated for feasibility in community pharmacies. Participants will be in one of two groups: intensive or abbreviated. Smoking abstinence rates, self-efficacy and overall satisfaction will be compared. Additionally, a cost-effectiveness analysis will be executed to determine the feasibility of customized smoking cessation programs in community pharmacies across Newfoundland and Labrador.

DETAILED DESCRIPTION:
One in five deaths in Canada is linked to smoking. It kills up to 50% of its users and over 7 million people each year. Smoking is also a risk factor for several harmful health consequences that affect the quality of life of those who smoke. It also results in substantial economic costs to society.

Newfoundland and Labrador (NL) has the highest smoking prevalence of Canadian provinces; approximately 18.5% of Newfoundlanders smoke on a daily or occasional basis compared to the national average of 13.0%. The Conference Board of Canada reported this year that smoking costs the local NL economy approximately $135 million per year in direct healthcare costs and $53 million in indirect costs, for a total of $188 million.

According to the CAN-ADAPTT Smoking Cessation Clinical Practice Guideline, several intensive counseling interventions are the most effective for smoking cessation. Offering a combination of counseling and pharmacotherapy increases the likelihood that a person will try to quit by 40-60%. Using this evidence, Memorial University's School of Pharmacy recently established a smoking cessation program at the Medication Therapy Services (MTS) Clinic. The program involves in-depth pharmacist consultation, which includes pharmacotherapy and multiple follow-up counseling sessions.

The investigators propose to test the effectiveness of an intensive and abbreviated smoking cessation program (SCP) delivered by trained pharmacists at the MTS Clinic. They hope that findings from this study will inform stakeholders of the value of the program and of the pharmacists' role. If the program is determined to be effective it could be instrumental in applying smoking cessation programs in community pharmacies across the province, including rural and remote locations.

To date there are only a small number of studies that use the randomized, controlled trial design to evaluate the effectiveness of pharmacist delivered interventions. In addition, data is lacking on the perspective of and satisfaction with smoking cessation services from the eyes of someone who participates in the program. Therefore, this study proposes to execute a randomized control trial to determine the effectiveness of a pharmacist-led smoking cessation program. Cost-effectiveness and a qualitative assessment of participant's journey to quit smoking will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults including anyone 19 or older who wish to make a change in their smoking.

Exclusion Criteria:

* People who do not smoke

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Abstinence Rate | 6 months
  To compare abstinence rates among participants who make a quit attempt, receiving either an intensive or abbreviated version of a pharmacist delivered smoking cessation program vs. those who receive usual care.

SECONDARY OUTCOMES:
Abstinence Rate | 3 months
  To compare abstinence rates among participants who make a quit attempt, receiving either an intensive or abbreviated version of a pharmacist delivered smoking cessation program vs. those who receive usual care.
Quit Attempts | 3 months
  To compare the number of quit attempts (defined as 24 hours or more of not smoking) and smoking reduction between each group.
Quit Attempts | 6 months
  To compare the number of quit attempts (defined as 24 hours or more of not smoking) and smoking reduction between each group.
Change in baseline quality of life measured using the European Quality of Life-5 Dimensions 3 Levels (EQ-5D-3L) survey | 0 and 6 months
  To compare the change in quality of life between each group.
Change in baseline self-efficacy using a self efficacy survey | 0 and 6 months
  To compare the change in self-efficacy between each group.
Satisfaction survey | 6 months
  A measure of the satisfaction of participants with receiving a pharmacist delivered smoking cessation program, or quitting using usual care.
Cost-effectiveness using an estimate an incremental cost per quality adjusted life year (QALY) gained | 6 months
  To assess the cost-effectiveness of an intensive, and abbreviated, pharmacist delivered smoking cessation support program vs. usual care. The cost of delivering each service will be combined with the outcome of each to estimate an incremental cost per quality adjusted life year (QALY) gained.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Genge, Principal Investigator — Memorial University, School of Pharmacy; Leslie Phillips, Principal Investigator — Memorial University, School of Pharmacy
Locations (1):
- School of Pharmacy, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] The World Health Organization: Tobacco (http://www.who.int/mediacentre/factsheets/fs339/en/)
- [Background] Dobrescu, Bhandari, Sutherland and Dinh (2017). The Costs of Tobacco Use in Canada, 2012. The Conference Board of Canada. Retrieved from http://www.conferenceboard.ca/e-library/abstract.aspx?did=9185
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Background] Reid JL, Hammond D, Rynard VL, Madill CL, Burkhalter R. Tobacco Use in Canada: Patterns and Trends, 2017 Edition. Waterloo, ON: Propel Centre for Population Health Impact, University of Waterloo.
- [Background] Government of Newfoundland and Labrador. (2017). The way forward: Realizing our potential. Retrieved from http://thewayforward.gov.nl.ca/documents/Realizing_our_potential.pdf
- [Background] Locke, Wade. (2017). State of N.L. Economy: From Bad to Worse. Presentation by Department of Economics, Memorial University.
- [Background] Gagnon-Arpin, Isabelle, Alexandru Dobrescu, Greg Sutherland, Carole Stonebridge, and Thy Dinh. The Value of Expanded Pharmacy Services in Canada. Ottawa: The Conference Board of Canada, 2017.
- [Background] CAN-ADAPTT. (2011). Canadian Smoking Cessation Clinical Practice Guideline. Toronto, Canada: Canadian Action Network for the Advancement, Dissemination and Adoption of Practice-informed Tobacco Treatment, Centre for Addiction and Mental Health.
- [Background] Aveyard P, Begh R, Parsons A, West R. Brief opportunistic smoking cessation interventions: a systematic review and meta-analysis to compare advice to quit and offer of assistance. Addiction. 2012 Jun;107(6):1066-73. doi: 10.1111/j.1360-0443.2011.03770.x. Epub 2012 Feb 28. PMID 22175545
- [Background] Canadian Association of Occupational Therapists; Canadian Association of Social Workers; Canadian Dental Association; Canadian Medical Association; Canadian Nurses Association; Canadian Pharmacists Association; Canadian Physiotherapy Association; Canadian Psychological Association; Canadian Society of Respiratory Therapists. Tobacco: the role of health professionals in smoking cessation. Joint statement. J Can Dent Assoc. 2001 Mar;67(3):134-5. No abstract available. PMID 11315390
- [Background] Canadian Pharmacists Association. Professional Development-QUIT program. https://www.pharmacists.ca/education-practice-resources/professional-development/quit/
- [Background] Newfoundland and Labrador Pharmacy Board. Prescribing by Pharmacists Standards of Pharmacy Practice. http://www.nlpb.ca/media/SOPP-Prescribing-by-Pharmacists-Aug2015-revFeb2016.pdf
- [Background] Fai SC, Yen GK, Malik N. Quit rates at 6 months in a pharmacist-led smoking cessation service in Malaysia. Can Pharm J (Ott). 2016 Sep;149(5):303-312. doi: 10.1177/1715163516662894. Epub 2016 Aug 9. PMID 27708676
- [Background] Bock BC, Hudmon KS, Christian J, Graham AL, Bock FR. A tailored intervention to support pharmacy-based counseling for smoking cessation. Nicotine Tob Res. 2010 Mar;12(3):217-25. doi: 10.1093/ntr/ntp197. Epub 2010 Jan 25. PMID 20100808
- [Background] Saba M, Diep J, Saini B, Dhippayom T. Meta-analysis of the effectiveness of smoking cessation interventions in community pharmacy. J Clin Pharm Ther. 2014 Jun;39(3):240-7. doi: 10.1111/jcpt.12131. Epub 2014 Jan 13. PMID 24749899
- [Background] Dent LA, Harris KJ, Noonan CW. Randomized trial assessing the effectiveness of a pharmacist-delivered program for smoking cessation. Ann Pharmacother. 2009 Feb;43(2):194-201. doi: 10.1345/aph.1L556. Epub 2009 Feb 3. PMID 19193572
- [Background] Zillich AJ, Ryan M, Adams A, Yeager B, Farris K. Effectiveness of a pharmacist-based smoking-cessation program and its impact on quality of life. Pharmacotherapy. 2002 Jun;22(6):759-65. doi: 10.1592/phco.22.9.759.34073. PMID 12066966
- [Background] Maguire TA, McElnay JC, Drummond A. A randomized controlled trial of a smoking cessation intervention based in community pharmacies. Addiction. 2001 Feb;96(2):325-31. doi: 10.1046/j.1360-0443.2001.96232516.x. PMID 11182878
- [Background] Kennedy DT, Giles JT, Chang ZG, Small RE, Edwards JH. Results of a smoking cessation clinic in community pharmacy practice. J Am Pharm Assoc (Wash). 2002 Jan-Feb;42(1):51-6. doi: 10.1331/108658002763538071. PMID 11833517
- [Background] Vial RJ, Jones TE, Ruffin RE, Gilbert AL. Smoking cessation program using nicotine patches: linking hospital to the community. J Pharm Pract Res. 2002;32:57-62.
- [Background] Smith MD, McGhan WF, Lauger G. Pharmacist counseling and outcomes of smoking cessation. Am Pharm. 1995 Aug;NS35(8):20-9; 32. doi: 10.1016/s0160-3450(15)30095-7. PMID 7677052
- [Background] Crealey GE, McElnay JC, Maguire TA, O'Neill C. Costs and effects associated with a community pharmacy-based smoking-cessation programme. Pharmacoeconomics. 1998 Sep;14(3):323-33. doi: 10.2165/00019053-199814030-00008. PMID 10186470
- [Background] McGhan WF, Smith MD. Pharmacoeconomic analysis of smoking-cessation interventions. Am J Health Syst Pharm. 1996 Jan 1;53(1):45-52. doi: 10.1093/ajhp/53.1.45. PMID 8719289
- [Background] Brown TJ, Todd A, O'Malley C, Moore HJ, Husband AK, Bambra C, Kasim A, Sniehotta FF, Steed L, Smith S, Nield L, Summerbell CD. Community pharmacy-delivered interventions for public health priorities: a systematic review of interventions for alcohol reduction, smoking cessation and weight management, including meta-analysis for smoking cessation. BMJ Open. 2016 Feb 29;6(2):e009828. doi: 10.1136/bmjopen-2015-009828. PMID 26928025
- [Background] Thavorn K, Chaiyakunapruk N. A cost-effectiveness analysis of a community pharmacist-based smoking cessation programme in Thailand. Tob Control. 2008 Jun;17(3):177-82. doi: 10.1136/tc.2007.022368. Epub 2008 Feb 19. PMID 18285385
- [Background] Tran MT, Holdford DA, Kennedy DT, Small RE. Modeling the cost-effectiveness of a smoking-cessation program in a community pharmacy practice. Pharmacotherapy. 2002 Dec;22(12):1623-31. doi: 10.1592/phco.22.17.1623.34118. PMID 12495172